CLINICAL TRIAL: NCT04709302
Title: COVID-19 and Its Effects on Endothelium in HIV-Positive Patients in Sub-Saharan Africa: Cardiometabolic Risk, Thrombosis and Vascular Function
Brief Title: Effects of COVID-19 on Endothelium in HIV-Positive Patients in Sub-Saharan Africa
Acronym: ENDOCOVID
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Graz (Other)
Collaborators: University of Olso (Unknown); Kristiania University College (Other); Walter Sisulu University (Other); Lagos State University (Other); Management Sciences for Health (Other)
Responsible Party: Sponsor
Other Study IDs: ENDOCOVID
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Hiv; ART
MeSH Terms: conditions — COVID-19; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive, HIV-positive with ART: Patients tested positive for SARS-CoV-2 Patients tested positive for HIV who are on ART
  Interventions: Biological: COVID-19; Biological: HIV; Drug: ART
- COVID-19 positive, HIV-positive without ART: Patients tested positive for SARS-CoV-2 Patients tested positive for HIV ART naive group
  Interventions: Biological: COVID-19; Biological: HIV
- COVID-19 positive, HIV-negative: Patients tested positive for SARS-CoV-2 Patients tested positive for HIV ART naive group
  Interventions: Biological: COVID-19

INTERVENTIONS:
Biological: COVID-19 — Patients diagnosed with a COVID-19 infection
  Other Names: SARS-CoV-2 positive
Biological: HIV — Patients diagnosed HIV-positive
  Groups: COVID-19 positive, HIV-positive with ART; COVID-19 positive, HIV-positive without ART
Drug: ART — Patients on ART
  Groups: COVID-19 positive, HIV-positive with ART

SUMMARY:
Background: Coronavirus disease 2019 (COVID-19) has affected almost every country in the world, especially in terms of health system capacity and economic burden. People from sub-Saharan Africa (SSA) often face interaction between human immunodeficiency virus (HIV) infection and non-communicable diseases such as cardiovascular disease. Role of HIV infection and anti-retroviral treatment (ART) in altered cardiovascular risk is questionable and there is still need to further carry out research in this field. However, thus far it is unclear, what impact the COVID-19 co-infection in people living with HIV (PLHIV), with or without therapy will have. The ENDOCOVID project aims to investigate whether and how HIV-infection in COVID-19 patients modulates the time course of the disease, alters cardiovascular risk, and changes vascular endothelial function and coagulation parameters/ thrombosis risk.

Methods: In this long-term study, cardiovascular research on PLHIV with or without ART with COVID-19 and HIV-negative with COVID-19 will be carried out via clinical and biochemical measurements for cardiovascular risk factors and biomarkers of cardiovascular disease (CVD). Vascular and endothelial function will be measured by brachial artery flow-mediated dilatation (FMD), carotid intima-media thickness (IMT) assessments, and retinal blood vessel analyses, along with vascular endothelial biomarkers and coagualation markers. The correlation between HIV-infection in COVID-19 PLHIV with or without ART and its role in enhancement of cardiovascular risk and endothelial dysfunction will be assessed. Potential changes in these endpoints by COVID-19 will be followed for 4 weeks across the three groups (PLHIVwith or without ART and HIV negatives).

Impact of project: The ENDOCOVID project aims to evaluate in the long-term the cardiovascular risk and vascular endothelial function in PLHIV thus revealing an important transitional cardiovascular phenotype in COVID-19.

DETAILED DESCRIPTION:
Background:

SARS-CoV-2 has affected almost every country worldwide with regard to health system capacities and economic burden, so far. The typical clinical presentations of COVID-19 are fever, sore through, cough, dyspnea, abdominal pain and diarrhea. Approximately 15% of patients with COVID-19 must be hospitalized and 5% are critically ill, and often develop acute respiratory distress syndrome and need to be admitted to intensive care units. Risk of severe disease increases with age, male sex, and with co-morbidities such as chronic lung disease, CVDs, and diabetes. COVID-19 can also affect the nervous systems and cause loss of smell or taste sensation.

Populations in SSA are increasingly facing a double burden of disease involving the interaction between HIV-AIDS and non-communicable diseases such as CVDs. In general, vascular endothelial function can be regarded as a marker of the net harmful effects of cardiovascular risk factors on the vascular wall. HIV- infected patients have premature atherosclerosis and increased risk of ischemic heart disease. The cardiovascular risk represented by HIV-infection is moreover affected by anti-retroviral treatment (ART). ART may, among other effects, prompt dyslipidaemic and metabolic changes in patients over to systemic immune activation, stimulation of endothelial inflammation and atherosclerosis. However, a recent meta-analysis showed that evidence for - and against - a role for ART in the development of CVDs remains unconvincing and that more research is necessary.

With the current COVID-19 pandemic, which has also spread across Africa, another burden is added. However, thus far it is unclear, what effect the additional COVID-19 co-infection in people with HIV (PLHIV) will have as there are no data yet on how HIV/AIDS a prevalent diseases SSA, will affect COVID-19 infection rates or outcomes. Currently, there is no proof for a higher COVID -19 infection rate in PLHIV compared to HIV-negatives. However, there is a possibility that HIV infection may have an influence on the course of infection. PLHIV who are on ART with a normal CD4 T-cell count and suppressed viral load should not be at an increased risk of severe disease. On the other hand, this theoretically positive situation could be counterbalanced by recent evidence that ART could also have effects on COVID-19. Furthermore, HIV-infected patients may additionally suffer from co-morbidities, which could pose a greater risk of COVID-19 infection. Currently, there is no data available about COVID-19 infection in PLHIV in SSA reflecting who in particular is at high risk for infections, complications and fatal outcomes. As COVID-19 associated multisystem inflammation, and the way organ damage caused by COVID-19 occurring in patients with COVID-19 is still incompletely understood, and current treatment options are limited. There is therefore an urgent need to better understand the risk of severe and fatal COVID-19 outcomes, especially in PLHIV (+/- ART).

A severe course of COVID-19 can cause the development of COVID-19-associated coagulopathy, with features of both disseminated intravascular coagulation and thrombotic microangiopathy, resulting in widespread microvascular thrombosis that may involve consumption of coagulation factors and the liver. There seems to be a causal relationship with the inflammatory and reparative processes involving diffuse alveolar damage (DAD), because thrombi are frequently detected in small pulmonary arteries, most presumed secondary to endothelial damage. The damage of endothelium could be due to the direct viral infection of the endothelial cells, which express ACE-2 receptors, or to a host response. Besides, the alveolar fibrin deposition in DAD may affect the local homeostasis between fibrinolysis and coagulation. Alveolar and endothelial damage of smaller vessels may be followed by microvascular pulmonary thrombosis, which could then extend to larger vessels. Additionally, elevated D-dimer has been observed in patients with COVID-19. It is known that inceased D-dimer is associated with acute pulmonary emboli (APE), deep venous thrombosis (DVT), cancer, peripheral vascular disease, inflammatory diseases and pregnancy. It has been found that patients with COVID-19, including those not on respirators but bedconfined, develop DVT and APE much earlier than expected. Even with usage of prophylactic anticoagulation, autopsy has shown that deaths in COVID-19 may be caused by the thrombosis in segmental and subsegmental pulmonary arterial vessels. ENDOCOVID project aims to evaluate the degree to which COVID-19 induced inflammation contributes to endothelial function and coagulation changes and cardiometabolic risk in PLHIV (+/-ART). Endothelial function will be evaluated non-invasively via FMD and blood asymmetric dimethyl arginine (ADMA).

Problem statement HIV infection is a burden for the cardiovascular system but coinfection of HIV and SARS-CoV-2 in SSA population could be a very big load and could lead to higher menace of cardiovascular health. However, the potential of risk in this population, including early vascular and endothelial changes, is yet unclear. Given the ongoing global pandemic, epidemiological studies to address this knowledge gap is necessary. The aim of this study is to evaluate cardiovascular risk in HIV and COVID-19 populations, which also would allow assessment of current - and future - cardiovascular risk, via vascular endothelial function measurements. The ENDOCOVID project has been designed to give an evaluation of cardiovascular risk in PLHIV and COVID-19 living in SAA. ENDOCOVID builds up on the EndoAfrica study, which is currently being carried out in SSA.

Aim and objectives The general aim of the ENDOCOVID project is to identify whether and how HIV-infection with or without ART in COVID-19 patients relates to the time course of the disease, alters cardiovascular risk, and changes vascular endothelial structure and function in adults living in the SSA.

Three groups of participants will take part in this project:

1. PLHIV without ART but with COVID-19
2. PLHIV with ART and COVID-19
3. HIV-negative patients with COVID-19, sex- /age matched

The following objectives will be investigated:

1. Evaluation of the prevalence of COVID-19 in PLHIV (with or without ART) admitted to clinics in South Africa and Nigeria because of COVID-19.
2. Assessment of the incidence of acute respiratory distress syndrome, admission to ICU, fatal course of disease (30-days mortality), and thromboembolic events in hospitalized patients included in the study.
3. Evaluation of the influence of ART on severity of COVID-19 in PLHIV (with or without ART) as well as clinical presentation, changes of endothelial/vascular function and biomarkers.
4. Evaluation of the effects of COVID-19 on endothelial/vascular function, thrombotic factors, and oro-naso sensory alterations over infection and after recovery.
5. Correlation of hospitalization and mortality of COVID-19 infected PLHIV(with or without ART) and HIV negatives with co-morbidity incidence;
6. Assessment of the incidence of obesity and insulin resistance in the 3 groups.

ELIGIBILITY:
Inclusion criteria:

* PLHIV without antiretroviral therapy but with COVID-19 infection
* PLHIV with antiretroviral therapy and COVID-19 infection
* HIV-negative patients, sex- and age matched, infected with COVID-19;
* older than 18 years

Exclusion criteria:

* Those with known co-infections such as hepatitis B and C
* with a viral load of HIV RNA >1000 copies/ml under ART or with advanced symptoms of AIDS
* negative for SARS-CoV-2 RNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the ENDOCOVID study population are patients with COVID-19, who at the same time are infected with HIV (with or without ART), or are HIV negative. Some may be admitted in the ICU. For inclusion into the study, participants must be positive for SARS-CoV-2 RNA and 18 years or older. Participants will be excluded from the study if they are less than 3 months post-partum and those with other co-infections than HIV such as tuberculosis Participants fulfilling the criteria will be invited into the study and asked to provide written informed consent.
Sampling Method: Probability Sample
Enrollment: 342 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients developing Acute Respiratory Distress Syndrome | through study completion, up to 3 months
  Comparison of all three groups, recorded for each patient
Number of ICU admissions | through study completion, up to 3 months
  Comparison of all three groups, recorded for each patient
Number of Deaths | through study completion, up to 3 months
  Comparison of all three groups

SECONDARY OUTCOMES:
Cardiometabolic Status: ADMA | through study completion, an average of 3 months
  Asymmetric dimethylarginine (ADMA) as marker for endothelial function (from blood sample) measured via commercially available ELISA kits
Cardiometabolic Status: Cholesterol | through study completion, an average of 3 months
  To assess the lipid profile, cholesterol levels will be assessed via blood samples in a routine laboratory
Cardiometabolic Status: Triglycerides | through study completion, an average of 3 months
  To assess the lipid profile, triglyceride concentrations will be assessed via blood samples in a routine laboratory
Cardiometabolic Status: HDL cholesterol | through study completion, an average of 3 months
  To assess the lipid profile, HDL cholesterol concentrations will be assessed via blood samples in a routine laboratory
Cardiometabolic Status: LDL cholesterol | through study completion, an average of 3 months
  To assess the lipid profile, LDL cholesterol concentrations will be assessed via blood samples in a routine laboratory
Cardiometabolic Status: Glucose | through study completion, an average of 3 months
  Assessed via blood samples in a routine laboratory
Cardiometabolic Status: Glycated Hemoglobin | through study completion, an average of 3 months
  HbA1c as marker for diabetes, assessed via blood samples in a routine laboratory
Cardiometabolic Status: hs-CRP | through study completion, an average of 3 months
  high sensitivity CRP as inflammatory marker, assessed via blood samples in a routine laboratory
Endothelial function and vascular changes: FMD | through study completion, an average of 3 months
  Assessed non-invasively using ultrasound in the brachial artery (flow mediated dilatation)
Endothelial function and vascular changes: PWV | through study completion, an average of 3 months
  PWV, a marker of aortic stiffness, is most commonly measured as the time it takes a pulse wave to travel from the carotid to the femoral arteries divided by the distance multiplied by 0.8. PWV can be measured by several devices. The non-invasive Vicorder device has been shown to have good reproducibility - even when the assessor has limited experience in its usage - and the results obtained reflect those obtained via invasive central blood pressure measurements and those of SphygmoCor device.
Endothelial function and vascular changes: Retinal microvasculature analysis | through study completion, an average of 3 months
  A non-mydriatic, hand-held, portable digital retinal camera (Optomed Aurora, Optomed Oy, Oulu, Finland) will be used for collecting retinal images. Dimensions of vessels and microvascular state will be analyzed offline with the semi-automated MONA REVA software (VITO, Belgium).
Endothelial function and vascular changes: IMT | through study completion, an average of 3 months
  Intima media thickness is assessed via ultrasound in the carotid artery
Coagulatory Parameters: D-dimer | through study completion, an average of 3 months
  increased D-Dimer as marker for pulmonary embolism in a routine laboratory
Coagulatory Parameters: CAT | through study completion, an average of 3 months
  Calibrated automated thrombography as thrombosis marker (Thrombinoscope BV)
Coagulatory Parameters: TF | through study completion, an average of 3 months
  Tissue factor (TF) measured via triggered thromboelastometry (TEM) coagulation analyzer (ROTEM05)

CONTACTS AND LOCATIONS:
Overall Officials: Nandu Goswami, Dr PhD, Principal Investigator — Medical University of Graz
Locations (3):
- Nigeria (2):
  - University of Ilorin Teaching Hospital, Ilorin, Kwara State
  - Lagos Stae University Teaching Hospital Ikeja, Lagos
- Walter Sisulu University, Mthatha, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goswami N, Fredriksen PM, Lundin KEA, Agu C, Elias SO, Motaung KS, Brix B, Cvirn G, Sourij H, Stelzl E, Kessler HH, Salon A, Nkeh-Chungag B. COVID-19 and its effects on endothelium in HIV-positive patients in sub-Saharan Africa: Cardiometabolic risk, thrombosis and vascular function (ENDOCOVID STUDY). BMC Infect Dis. 2021 Jul 31;21(1):719. doi: 10.1186/s12879-021-06426-8. PMID 34332551